CLINICAL TRIAL: NCT06517056
Title: Objective Dynamic and 3D Knee Assessment Medical Device to Improve Recovery and Accelerate Return to Readiness in Service Members With Knee Pain
Brief Title: Emovi 3D Knee Assessment Device Intervention for Operational Readiness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: WAMC.2024.0053
Record Dates: First submitted 2024-06-10; First posted 2024-07-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Patellofemoral Pain; Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain; Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: The study design is with 1:1 treatment arms: 1) KneeKG informed cared or 2) usual care without any information from the KneeKG
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention: Knee KG informed physical therapy (Experimental): Participants in this group will receive care guided by the impairments identified with the KneeKG. The KneeKG exam results in recommended exercises that target the specific biomechanical impairments identified. The exercises and dose given to the participant will be based on what the KneeKG device recommends after the exam. The participant will be seen twice a week for 4 weeks.
  Interventions: Device: Emovi Knee Kinesiography
- Control: Standard of care physical therapy (No Intervention): Participants in this arm will have their KneeKG data captured, but this information will not be provided to the physical therapist to inform their care. Instead, physical therapists will deliver care as they normally do in routine clinical practice. The participant will be seen twice a week for 4 weeks.

INTERVENTIONS:
Device: Emovi Knee Kinesiography — All participants will receive a KneeKG exam. This device will capture three-dimensional knee kinematics for a participant's knee, using the KneeKG system. Therapists will use these reports and suggested exercises to guide their care for participants in the Intervention group.
  Other Names: KneeKG
  Arms: Intervention: Knee KG informed physical therapy

SUMMARY:
This is a randomized clinical trial investigating the use of the Emovi Knee Kinesiography information in the treatment of anterior knee pain in physical therapy.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness of using a 3D medical assessment device versus usual care to help guide clinical decisions about the management of PFP. The objective is to determine if gathering objective biomechanical data from a three-dimensional (3D) motion capture device leads to more precise and optimal care, ultimately improving physical function and other outcomes compared to participants who receive routine care that is not guided by information from this device.

Participants will be recruited from primary care and physical therapy clinics at participating sites. Authorized study personnel will search electronic medical records (Genesis) to identify potential study participants diagnosed with knee pain.

After consent and enrollment, participants will complete baseline measures and then receive a Knee Kinesiography exam. The participant will be entered into the KneeKG system using a unique participant identifier. After the knee kinesiography exam with the KneeKG, participants will be randomized 1:1 into one of two different treatment arms: 1) KneeKG informed care or 2) usual care without any information from the KneeKG.

Knee mechanics during gait is assessed with a Knee Kinesiography exam. The participant will walk for 5 minutes on a commercial treadmill at their comfortable speed. Three-dimensional (3D) knee kinematics are captured on each leg using the KneeKG system (Emovi, Canada). With this validated FDA cleared medical device, there is an accurate quantification of specific knee biomechanical markers during gait in a clinical setting. There will be two 45-second trials to electronically capture the data which is immediately accessible through automatic reports. Biomechanical markers captured include but are not limited to varus/valgus alignment at stance, varus/valgus alignment at heel strike, knee flexion angle at heel strike, total knee excursion in sagittal plane, tibial rotation at heel strike and throughout gait cycle. The entire procedure will take approximately 15-20 minutes. This procedure will occur at baseline and also again at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Active Duty Service Member stationed at Fort Liberty and Schofield Barracks
* Diagnosis of patellofemoral pain (ICD-10 codes: M25.2 (pain in unspecified knee), M25.561 (pain in right knee), and M25.562 (pain in left knee)

Exclusion Criteria:

* Pregnancy
* Known to be leaving that duty station within next 3 months
* Concurrent lower limb injuries (examples include but are not limited to ankle sprain or HS strain)
* Previous knee surgery
* History of traumatic knee injury, such as a ligament tear or meniscal tear
* Presence of rheumatoid or neurological disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function | 12 weeks
  PROMIS asks patients about their functional ability, and symptoms. This tool is designed as a health-focused rather than a disease-focused measurement system. The primary outcome measure will focus on the the Physical Function domains since PFPS is known to limit function during daily and sports & recreation activities. This is an adaptive questionnaire that is taken in RedCap and contains up to 166 questions that will not all be asked, scored 1-5 on a Likert scale based on limits of function.
  The primary outcome is the between-group difference in PROMIS Physical Function T-score at 3 months. A linear mixed effects model will be used to analyze the between-group differences across the various time points (repeated measures).

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference | 12 weeks
  This PROMIS tool focuses on pain interference in daily life. This questionnaire is adaptive taken in RedCap and contains up to 41 questions that will not all be asked. It is scored on a 5 point Likert scale based on limitation due to pain.
Anterior Knee Pain Scale (AKPS) | 12 weeks
  The Anterior Knee Pain Scale is a 13-item more specific questionnaire related to PF pain which will allow to assess pain and symptoms during specific loading-activities. The 13 items on the scale are used to assess subjective symptoms and functional restrictions. A score can have a minimum of 0 points or a maximum of 100 points. Athletes would receive a score of 100 if they showed no signs of anterior knee pain.
Self-Reported Readiness to Return to Duty | 12 weeks
  The Self-Reported Readiness to Return to Duty questionnaire consists of three questions to assess perceived readiness to return to duty
Total Lost Duty Days | 12 weeks
  Tracking the amount of duty days a soldier missed while enrolled in protocol.
Provider Satisfaction | 12 weeks
  A provider satisfaction survey will be used to measure patient satisfaction with quality of physical therapy care.

CONTACTS AND LOCATIONS:
Overall Officials: Don L Goss, DPT, PhD, Principal Investigator — Womack Army Medical Center
Locations (2):
- United States (2):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Womack Army Medical Center, Fort Liberty, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT06517056/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT06517056/ICF_001.pdf